CLINICAL TRIAL: NCT00601445
Title: Homeostatic Sleep Regulation in Older Persons
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute on Aging (NIA) (NIH)
Collaborators: Brigham and Women's Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: AG0090; P01-AG009975 - Project 4; P01AG009975 (NIH)
Record Dates: First submitted 2007-10-24; First posted 2008-01-28 (Estimated); Last update posted 2008-05-30 (Estimated); Status verified 2008-05

CONDITIONS: Healthy; Aging
Keywords: Changes in sleep with aging

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Behavioral: Amount of sleep and wake — 4 groups with different patterns of sleep and wake

SUMMARY:
The purpose of this study is to test the hypothesis that sleep homeostasis, also known as sleep pressure or sleep drive, is different in healthy older and younger individuals.

DETAILED DESCRIPTION:
This was an inpatient study of healthy individuals to determine whether homeostatic "sleep drive" effects on sleep change with healthy aging. Sleep, performance, and mood were studied on individuals sleeping different lengths of time and during wake periods of different durations.

ELIGIBILITY:
Inclusion Criteria:

* Ages 18-30 and 60-85 years
* Healthy

Exclusion Criteria:

* Any medications
* Sleep Disorder

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 58 (Estimated)
Dates: Start 1999-09; Study Completion 2004-03 (Actual)

PRIMARY OUTCOMES:
Total Sleep Time | During inpatient study

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth B Klerman, MD, PhD, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States